CLINICAL TRIAL: NCT03232333
Title: Effectiveness of MIRODERM® Biologic Wound Matrix in the Treatment of Hard-to-Heal Diabetic Foot Ulcers
Brief Title: MIRODERM H2H DFU Study
Acronym: H2H-DFU
Status: Completed | Type: Observational
Sponsor: Miromatrix Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016002
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Debridement waste
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MIRODERM: Biologic wound graft
  Interventions: Device: Biologic wound graft

INTERVENTIONS:
Device: Biologic wound graft — Diabetic foot ulcer will be treated by grafting with MIRODERM Biologic Wound Matrix
  Other Names: MIRODERM Biologic Wound Matrix treatment

SUMMARY:
This study will assess the ability of MIRODERM to heal difficult diabetic foot ulcers within 12 weeks of treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the number of successful complete wound closures within 12 weeks of treatment with MIRODERM Fenestrated Biological Wound Matrix. Some secondary objectives of this study include documenting the time course of wound healing and assessing changes in quality of life.

The primary cohort is individuals suffering from a diabetic foot ulcer that has not been healed in the last 3 months and after at least 2 attempts with an advanced biologic. Ulcer will be between 1 and 12 cm squared, less than 5 mm deep, full thickness, below the ankle, and with no exposed bone or tendon. Subjects will be 18 or older, have Type I or II diabetes with adequate vascular profusion. Subjects will be unable to participate if they have osteomyelitis, Charcot foot, a known collagen vascular disease, are on dialyses, are immunocompromised or have an HbA1c level equal to or great than 12%.

This is a single-arm study with no Independent Variables. Descriptive data to be collected will include demographics, pathology and medical history.

Outcome assessments:

* proportion of subjects with 100% epithelialization of wound
* SF-36
* Adverse events

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older at time of initial visit
* Have Type I or Type II diabetes
* Have a neuropathic diabetic foot ulcer with the following characteristics:

  * Is greater than 1 cm2 and less than or equal to 12 cm2
  * Has failed to close following at least 2 treatments with a biologic
  * Has been present for 90 days or longer
  * Does not show signs of infection
  * Is full thickness (Wagner Grade I or II)
  * Located distal to the malleolus
  * Depth of less than or equal to 5 mm
  * No exposed capsule, tendon or bone
  * No tunneling, undermining or sinus tracts
  * Not between the toes
* Be willing and able to maintain required off-loading of affected limb
* Be willing and able to perform necessary dressing changes
* Have at least one of the following:

  * An Ankle-brachial index (ABI) ≥ 0.8
  * TcPO2 of ≥ 30 mmHg
  * A toe pressure of ≥ 50 mmHg

Exclusion Criteria:

* Be pregnant or be planning to become pregnant during the study
* Have had a Chopart's Amputation (or higher)
* Have a history of bone cancer of the affected limb
* Be undergoing dialysis
* Have active osteomyelitis or be receiving treatment for osteomyelitis
* Be diagnosed with unstable Charcot Foot on the affected side
* Have an HbA1c level of ≥ 12% within the past 90 days
* Have another ulcer within 2 cm of the study ulcer
* Be immunocompromised or at risk of immunosuppression as determined by the treating investigator
* Have a known collagen vascular disease or connective tissue disease
* Have received treatment of the study ulcer with a skin substitute product or topical growth factor within the past 4 weeks
* Be participating in another medical research study
* Have a sensitivity to porcine material

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who have at least one small to moderately sized diabetic foot ulcer and have been undergoing extended and unsuccessful treatment, as defined by failure of the wound to completely close over the previous 3 months and after application of at least 2 biological products.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fridman, DPM, Principal Investigator — Foot Associates of New York; M Mason Macenski, PhD, Study Director — Miromatrix
Locations (9):
- United States (9):
  - ILD Research, Carlsbad, California
  - Bond Clinic / Clinical Reseach of Central Florida, Winter Haven, Florida
  - American Health Network, Avon, Indiana
  - Kansas City Institute of Podiatry, Overland Park, Kansas
  - St. Anthony's Wound Care Center, St Louis, Missouri
  - A Step Ahead Foot Care, Mount Vernon, New York
  - Gramercy Park Podiatry, New York, New York
  - Foot Associates of New York, New York, New York
  - Foot and Ankle Institute, St. George, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MIRODERM: Biologic wound graft: Diabetic foot ulcer was treated with MIRODERM Biologic Wound Matrix
Period: Overall Study
Arm/Group | MIRODERM
Started | 53
Completed | 38
Not Completed | 15
Not completed — Infection or Osteomyelitis | 9
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | MIRODERM
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 8 are hispanic
  Participants
    number analyzed (Participants) | 30
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 2
    Black or African American | 5
    White | 21
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 38
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.2 (6.3)
HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 7.8 (1.5)
Ankle Brachial Index [Mean (Standard Deviation); unit: Ratio] — The Ankle Bronchial Index (ABI) is the systolic blood pressure reading obtained at the ankle divided by the systolic blood pressure reading from an arm. An ABI of 0.9 or may indicate peripheral vascular insufficiency. An ABI ratio between 1.0 and 1.4 is normal
  Ratio | 1.02 (0.2)
Tobacco Use [Count of Participants; unit: Participants]
  None | 34
  < 1 pack/day | 3
  > 1 pack/day | 1
Alcohol Use [Count of Participants; unit: Participants]
  None | 28
  Occasional | 5
  Monthly | 3
  Weekly | 1
  Daily | 1
Wound Size Screening [Mean (Standard Deviation); unit: cm^2] | 3.5 (3.5)
Wound Size Treatment [Mean (Standard Deviation); unit: cm^2] | 3.5 (3.8)
Wound Age [Mean (Standard Deviation); unit: weeks] | 41.1 (27.2)
Prior Treatments [Median (Full Range); unit: Applications] | 2 [2 to 13]
Wound Location [Count of Participants; unit: Participants]
  Toes | 3
  Forefoot | 14
  Midfoot | 14
  Heel | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants
Description: Percentage of participants with healed ulcers within 12 weeks of treatment
Time Frame: 12 weeks
Population: Per protocol analysis
Measure: Number; unit: Percentage of participants with healed u
Arm/Group | MIRODERM
Number analyzed (Participants) | 38
Percentage of participants with healed u | 57.89

2. Other Pre Specified Outcome: MIRODERM Applications
Description: Frequency of MIRODERM applications prior to wound closing
Time Frame: 12 weeks
Population: Per protocol analysis
Measure: Median (Full Range); unit: Applications
Arm/Group | MIRODERM
Number analyzed (Participants) | 38
Applications | 2.0 [1 to 10]

3. Other Pre Specified Outcome: Time to Closure
Description: Measures the time from treatment to wound healing
Time Frame: 12 weeks
Population: Subjects who healed in 12 weeks or less
Measure: Mean (Full Range); unit: Weeks
Arm/Group | MIRODERM
Number analyzed (Participants) | 22
Weeks | 8.1 [2 to 12]

4. Other Pre Specified Outcome: Change in Patient's Wound Size
Description: Gives the mean area that the wound closed per week
Time Frame: 12 weeks
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: cm^2 per week
Arm/Group | MIRODERM
Number analyzed (Participants) | 38
cm^2 per week | 0.30 (0.28)

5. Other Pre Specified Outcome: Short Form F36 - Physical Component Summary Score
Description: Measure Description: The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Physical Function, Role Physical, Bodily Pain, and General health which assess aspects of physical health. These are used to make an overall physical health score, the Physical Component Summary score (PCS). The higher the score the better the subject's physical health. Range from 0-100.
Time Frame: Baseline (Pre-Procedure) and then at final follow-up (maximum 12 weeks)
Population: Subjects who's ulcer healed in 12 weeks or less two without appropriate data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIRODERM
Number analyzed (Participants) | 20
score on a scale
  Pre-procedure | 39.0 (16.7)
  Follow-up | 37.0 (25.6)
Statistical Analysis 1: Comparison: MIRODERM; Test type: Superiority; p = 0.71, t-test, 1 sided

6. Other Pre Specified Outcome: Short Form 36 - Mental Component Summary Score
Description: Measure Description: The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Vitality, Role Emotional, Social Functioning, and Mental health which assess aspects of Mental health. These are used to make an overall mental health score, the Mental Component Summary score (MCS). The higher the score the better the subject's mental health. Range from 0-100.
Time Frame: Baseline (Pre-Procedure) and then at final follow-up (maximum 12 weeks)
Population: Subjects who's wound healed in 12 weeks or less one without appropriate data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIRODERM
Number analyzed (Participants) | 21
score on a scale
  Pre-procedure | 71.0 (16.9)
  Follow-up | 71.9 (13.9)
Statistical Analysis 1: Comparison: MIRODERM; Test type: Superiority; p = 0.63, t-test, 1 sided

7. Other Pre Specified Outcome: Short Form - 36: Bodily Pain
Description: Measure Description: The Short-Form 36 (SF-36) is a general health assessment tool comprised of 8 sub-scales including Bodily Pain which assess aspects of physical pain. The higher the score the better the subject's physical health with respect to feeling pain. Range from 0-100.
Time Frame: Baseline (Pre-Procedure) and then at final follow-up (maximum 12 weeks)
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIRODERM
Number analyzed (Participants) | 21
score on a scale
  Pre-procedure | 57.5 (32.2)
  Follow-up | 61.9 (29.0)
Statistical Analysis 1: Comparison: MIRODERM; Test type: Superiority; p = .01, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | MIRODERM
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 2/53
Other Adverse Events (participants affected / at risk) | 11/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIRODERM (N=53)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIRODERM (N=53)
Cellulitis (Infections and infestations) | 4 (5)
Infection (Infections and infestations) | 2 (2)
Increase in wound size (Skin and subcutaneous tissue disorders) | 1 (1)
Wound abscess (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (3)

LIMITATIONS AND CAVEATS:
Not a randomized trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03232333/Prot_SAP_000.pdf